CLINICAL TRIAL: NCT00232960
Title: Postoperative Radiotherapy According to Molecular Analysis of Surgical Margins of Early Stages Oral and Oropharyngeal Squamous Cell Carcinomas: A Prospective Study
Brief Title: Postoperative Radiotherapy According to Molecular Analysis of Surgical Margins of Oral and Oropharyngeal SCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Tumor Study Group Head and Neck (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Marges-ORL
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Oral Cancer; Oropharynx Cancer
Keywords: oral and oropharynx carcinoma; surgery; postoperative radiotherapy; molecular analysis; microsatellite instability
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms; Microsatellite Instability

INTERVENTIONS:
Procedure: Radiotherapy 50 Gy

SUMMARY:
There is no consensus on the indication of postoperative radiotherapy for early stages oral and oropharyngeal squamous cell carcinoma with complete pathological resection and no neck node metastasis, but most of the institutions do not give any post-operative treatment. Loco-regional control rates range between 80-85% at five years. Surgical margins molecular analysis for microsatellite instability (MSI) marker could help to select the high-risk patients who should receive postoperative radiotherapy. We expect to include 120 patients in five years and have 60 informative tumors for MSI marker. Patients with positive molecular margins will receive postoperative radiotherapy (50 Gy). Patients with negative molecular margins will not receive radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Oral and oropharynx (exclusion vallecula) squamous cell carcinoma
* T1 or T2
* unique, untreated tumor
* N0 or nodes <3cm
* complete pathological resection
* no perineural spread, vascular emboli <5
* pN0 or <=2N+R-
* signed inform consent

Exclusion Criteria:

* Vallecula carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2005-10; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
loco-regional control | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Temam, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (4):
- France (4):
  - Centre Francois Baclesse, Caen
  - Hôpital de la Croix Rousse, Lyon
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif